CLINICAL TRIAL: NCT05543577
Title: Comparative Study of the Preparedness and Knowledge of Pharmacists Versus Intern Physician in the Current Monkeypox Outbreak
Brief Title: Assessing the Preparedness and Knowledge of Pharmacists in the Current Monkeypox Outbreak
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Asmaa Abdelfattah Elsayed, Assistant lecturer, Beni-Suef University
Other Study IDs: BeniSuefU2022
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Monkey Pox
MeSH Terms: conditions — Mpox, Monkeypox | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pharmacists: community, hospital and clinical pharmacists
  Interventions: Other: Questionnaire
- Medical interns: Medical interns of both sexes
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire

SUMMARY:
General objective: to measure the preparedness of pharmacists and medical interns about monkeypox

Specific objectives: to evaluate the level of knowledge among pharmacists and medical interns about monkeypox treatment and nature of disease

DETAILED DESCRIPTION:
Globally, the ongoing outbreak was declared as a public health emergency. After the first laboratory-confirmed case of monkeypox was reported in Singapore on May 2019, countries all over the world started to strengthen disease surveillance systems. One challenge in preventing monkeypox is a lack of knowledge, particularly among healthcare workers.

Study significance: to examine in detail the preparedness and the perception of pharmacists and medical interns about monkeypox and to evaluate the level of knowledge about monkeypox management and nature of disease.

ELIGIBILITY:
Inclusion Criteria:

- community, hospital and clinical pharmacists, Medical interns of both sexes

Exclusion Criteria:

* any other healthcare professional

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community, hospital and clinical pharmacists, Medical interns of both sexes and any age
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
the level of knowledge among pharmacists and medical interns about monkeypox treatment and nature of disease using an online Questionnaire | 2 months
  the level of knowledge among pharmacists and medical interns about monkeypox treatment and nature of disease using a validated questionnaire
Direct interviews with the pharmacists and medical interns to assess their knowledge and attitudes about diagnosing and dealing with the Monkeypox infected cases | 2 months
  Direct interviews with the pharmacists and medical interns to assess their knowledge and attitudes about diagnosing and dealing with the Monkeypox infected cases

CONTACTS AND LOCATIONS:
Overall Officials: Engy Wahsh, Ph.D., Study Director — 6october University
Locations (1):
- BeniSuefU, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No
only the PI will keep the data and have access to the questionnaire

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35888642/